CLINICAL TRIAL: NCT05072639
Title: Preoperative Guided Imagery in Patients Undergoing Urologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15989; NCI-2021-10906 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Urologic Cancer
Keywords: Meditation; Guided Imagery; Urologic-oncology Surgery; Anxiety reduction; Radical cystectomy; Radical nephrectomy; Partial nephrectomy; Radical prostatectomy
MeSH Terms: conditions — Urologic Neoplasms | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation (Experimental): Participants randomized to the meditation arm will receive an mp3 audio recording of the visual guided meditation will be sent an additional mp3 file specifically for the recovery phase of surgery. Participants will be asked to complete a series of pre-study questionnaires to determine their baseline anxiety, depression, stress, and quality of life scores. Subjects will then complete the same questionnaires at four additional time points: after 10 days of daily meditations, 1 day before their surgery, and day after discharge, and 4 weeks post-operation.
  Interventions: Behavioral: Guided Meditation
- Control group (No Intervention): Participants received standard of care, including the option to attend a free "Prepare for Surgery workshop". Participants will be asked to complete a series of pre-study questionnaires to determine their baseline anxiety, depression, stress, and quality of life scores. Subjects will then complete the same questionnaires at four additional time points: after 10 days of daily meditations, 1 day before their surgery, and day after discharge, and 4 weeks post-operation.

INTERVENTIONS:
Behavioral: Guided Meditation — 23 minute audio recording
  Other Names: Meditation
  Arms: Meditation

SUMMARY:
This is a prospective randomized controlled trial of patients undergoing major urologic-oncologic surgery at the University of California, San Francisco (UCSF) Medical Center and the Helen Diller Family Comprehensive Cancer Center. This clinical trial examines the effect of guided meditation before surgery on the levels of anxiety, stress, sleep disturbance, and quality of life among patients scheduled to undergo a major urologic surgery for cancer. A cancer diagnosis and the treatments associated with it can be very stressful for patients, leading to depression, sleep disturbances, and lower quality of life. Mind-body practices such as guided meditation have been used for thousands of years to reduce the effects of chronic stress and to improve quality of life. This clinical trial examines the effects of guided meditation on the stress, depression, and quality of life levels of patients undergoing urologic surgery for their cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effect of 14 days of preoperative guided visualization meditation on patients' anxiety undergoing major urologic-oncology surgery.

SECONDARY OBJECTIVES:

I. To determine the effect of preoperative guided visualization meditation on patients' depression, stress, and quality of life.

II. To examine the difference in Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) Survey question scores between the two study groups.

III. To determine the ability of patient to perform a daily 23 minute meditation.

IV. To examine the correlation between depression and emergency department (ED) visits and readmissions post-operations.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients listen to guided meditation over 23 minutes daily for two weeks before their standard of care surgery. Patients also complete surveys over 10-15 minutes at baseline, after 10 days, 1 day before standard of care surgery, the day after discharge, and then 4 weeks after surgery.

ARM 2: Patients complete surveys over 10-15 minutes at baseline, after 10 days, 1 day before standard of care surgery, the day after discharge, and then 4 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age.
* Patients undergoing radical cystectomy, radical or partial nephrectomy, or radical prostatectomy at the University of California, San Francisco (UCSF) Medical Center and the Helen Diller Family Comprehensive Cancer Center
* Access to an electronic device that can play mp3 recording and for survey completion
* At least a 2 week window from date of surgical booking to the scheduled surgery

Exclusion Criteria:

* Inability to consent for the study (ie, they have a surrogate decision maker).
* Non-English speaker (the meditations are only available in English)
* Patients scheduled for surgery less than 2 weeks away

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-03-25 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in scores on the State-Trait Anxiety Inventory (STAI) from baseline to day before surgery | Up to 4 weeks
  The Spielberger et. al STAI is a commonly used measure of trait and state anxiety . It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It has 20 items for assessing trait anxiety and 20 for state anxiety for a total of 40 items. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "1=Almost Never" to 4="Almost Always") with a maximum score range of 40-160 when all 40 items are administered Higher scores indicate greater anxiety. A two sample t-test will be used to compare the change between anxiety scores from baseline to the time point the day before surgery for the population as a whole and then adjusted for by surgery type.

SECONDARY OUTCOMES:
Change in scores on the State-Trait Anxiety Inventory (STAI) over time | Up to 6 months
  The Spielberger et. al STAI is a commonly used measure of trait and state anxiety . It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It has 20 items for assessing trait anxiety and 20 for state anxiety for a total of 40 items. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "1=Almost Never" to 4="Almost Always") with a maximum score range of 40-160 when all 40 items are administered Higher scores indicate greater anxiety.
Change in scores on the Center for Epidemiologic Depression Scale (CESD) over time | Up to 6 months
  The Center for Epidemiological Studies-Depression (CESD) is a 20-item measure that asks caregivers to rate how often over the past week participants experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Change in scores on the Perceived Stress Scale (PSS) over time | Up to 6 months
  The PSS is a 10-item questionnaire which asks participants about feelings and thoughts during the last month. In each case, respondents are asked how often participants felt a certain way. Scores of each item ranging from 0 = "Never" to 4 = "Very Often" for a total score range of 0 to 40. Scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to 4 of the 10 positively stated items and scores are calculated by summing the total. Higher scores indicate higher degree of perceived stress.
Change in scores on the National Comprehensive Cancer Network (NCCN) Distress Thermometer over time | Up to 6 months
  The NCCN Distress Thermometer is a single item screening tool among cancer care providers. which measures distress by asking participants to report their level of distress in the past week on a 0 to 10 scale, with a score of 0='No distress' and 10='Extreme Distress'.
Change in scores on the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) for cancer patients (EORTC-QLQ-C30) - Functional Domains over time | Up to 6 months
  The functional domains measure the quality of life in Physical functioning, Role functioning, Emotional functioning, Cognitive functioning, Social functioning. Scores consists of responses to items with responses ranging from 1="Not at all" to 4="Very Much". The raw score is calculated by estimating the mean of the items that make up each domains with a resulting total range of 1 - 4. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score for the functional domains represents a high level of functioning
Change in scores on the EORTC-QLQ-C30 Global Health Status over time | Up to 6 months
  The global health status score consists of responses to two items with responses ranging from 1="very poor" to 4="excellent". The raw score is calculated by estimating the mean of the two items that make up the global health scale with a resulting total range of 1-7. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score for the global health status represents a higher quality of life.
Change in scores on the EORTC-QLQ-C30 - Symptoms over time | Up to 6 months
  The Pain score consists of responses to two items with responses ranging from 1="Not at all" to 4="Very Much". The raw score is calculated by estimating the mean of the two items that make up the pain scale with a resulting total range of 1-4. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score for the pain scale / item represents a high level of symptomatology / problems.
Mean scores on the Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) Survey | Up to 6 months
  HCAHPS is a 29-item survey for measuring patients' perceptions of their hospital experience. The questions address participants recent hospital stay and contain 19 core questions about critical aspects of patients' hospital experiences (communication with nurses and doctors, the responsiveness of hospital staff, the cleanliness and quietness of the hospital environment, communication about medicines, discharge information, overall rating of hospital, and would patients recommend the hospital). The survey also includes 3 items to direct patients to relevant questions, five items to adjust for the mix of patients across hospitals, and 2 items that support Congressionally-mandated reports. Total scores are calculated by summing the items in each domain with higher scores indicating a greater overall satisfaction. A comparison of mean scores of HCAHPS survey questions between the two study groups using a two sample t-test.
Proportion of participants who completed daily meditation | Up to 6 months
  Participants in the intervention arm will receive an automated text message once a week before their surgery to remind them of the daily meditation routine. Participants will then be asked to report how many days of completed meditations have been completed in the past week.
Percentage of emergency department (ED) visits at 4 weeks post-operative | 4 weeks
  The percentage of participants who visited the emergency department for an oncological related event within 4 weeks post surgery will be reported.
Rates of hospital re-admission rates at 4 weeks post operatively | 4 weeks
  The percentage of participants who were re-admitted to the hospital for an oncological related event within 4 weeks post surgery will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Sima Porten, MD,, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No